CLINICAL TRIAL: NCT00511342
Title: An Open-Label, Randomized, Single Center Trial in Healthy Young Women, to Evaluate the Effects of a Monophasic Combined Oral Contraceptive (COC) Containing 2.5 mg NOMAC and 1.5 mg E2 on Bone Mineral Density (BMD) Compared to a Monophasic COC Containing 0.150 mg Levonorgestrel and 0.030 mg Ethinyl Estradiol
Brief Title: Effects on Bone Mineral Density (BMD) of the Combined Oral Contraceptive NOMAC-E2 Compared to a COC Containing LNG/EE (292005)(P05765)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P05765; Organon Protocol No. 292005
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NOMAC-E2 (Experimental): Nomegestrol Acetate (NOMAC) and Estradiol (E2), 2.5 mg NOMAC and 1.5 mg E2 monophasic COC
  Interventions: Drug: NOMAC-E2
- LNG-EE (Active Comparator): Levonorgestrel (LNG) and Ethinyl Estradiol (EE), 0.150 mg LNG and 0.030 mg EE monophasic COC
  Interventions: Drug: LNG-EE

INTERVENTIONS:
Drug: NOMAC-E2 — Nomegestrol Acetate and Estradiol Tablets, 2.5 mg NOMAC and 1.5 mg E2 taken once daily from Day 1 of menstrual period up to and including Day 28 for 26 consecutive 28-day menstrual cycles (2 years).
  Other Names: SCH 900121
  Arms: NOMAC-E2
Drug: LNG-EE — Levonorgestrel and Ethinyl Estradiol Tablets, 0.150 mg Levonorgestrel and 0.030 mg Ethinyl Estradiol taken once daily from Day 1 of menstrual period up to and including Day 28 for 26 consecutive 28-day menstrual cycles (2 years).
  Other Names: SCH 900121
  Arms: LNG-EE

SUMMARY:
The primary purpose of this study is to evaluate the effects of the NOMAC-E2 combined oral contraceptive (COC) on bone mineral density (BMD).

ELIGIBILITY:
Inclusion criteria:

* Sexually active women, at risk for pregnancy and not planning to use condoms

during treatment;

* At least 20 but not older than 35 years of age at the time of screening;
* BMI = 17 and = 35;
* Good physical and mental health;
* Willing to give informed consent in writing;
* Willing to take part in the trial for two years.

Exclusion criteria:

* Family history of osteoporotic fracture below the age of 70;
* Postgastrectomy;
* History of eating disorder, viz. anorexia nervosa, bulimia;
* Endocrine disorder (including controlled diabetes, [para]thyroid disease, Cushing's disease);
* Rheumatoid arthritis;
* Significant scoliosis;
* Fasting parathyroid hormone (PTH) outside the reference range at screening;
* Fasting calcitonin outside the reference range at screening;
* Prolactin above the reference range (hyperprolactinemia) at screening;
* Fasting cholesterol and/or triglycerides above the reference range for age at screening (treatment with lipid lowering drugs not allowed);
* Engaging in vigorous exercise such as marathon, competitive swimming, triathlon;
* Smoking more than ten cigarettes/day;
* Use of more than two units of alcohol a day;
* Use of one or more of the following drugs:

  * gonadotropin releasing hormone (GnRH) analogues (also past use for more than six months at any time, or for any period of time less than six months ago is a contraindication);
  * systemic or inhaled administration of corticosteroids (also past use for more than one year, less than five years ago or any period of time in the past year is a contraindication);
  * thiazide diuretics;
  * thyroid hormone;
  * bisphosphonates;
  * calcium supplementation in combination with vitamin D supplementation/

calcitonin;

* ever treatment after childhood with fluorides;

  * Contraindications for contraceptive steroids
  * An abnormal cervical smear (i.e.: dysplasia, cervical intraepithelial neoplasia[CIN], squamous intraepithelial lesion [SIL], carcinoma in situ, invasive carcinoma) at screening;
  * Clinically relevant abnormal laboratory result at screening as judged by the investigator;
  * Use of an injectable hormonal method of contraception; within 6 months of an injection with a 3-month duration, within 4 months of an injection with a 2-month duration, within 2 months of an injection with a 1-month duration;
  * Within 12 months after a pregnancy prior to the start of trial medication;
  * Breastfeeding or within 12 months after stopping breastfeeding prior to the start of trial medication;
  * Present use or use within 2 months prior to the start of the trial medication of the following drugs: phenytoin, barbiturates, primidone, carbamazepine, oxcarbazepine, topiramate, felbamate, rifampicin, nelfinavir, ritonavir, griseofulvin, ketoconazole, sex steroids (other than pre- and post-treatment contraceptive method) and herbal remedies containing Hypericum perforatum (St John's Wort);
  * Administration of investigational drugs and/or participation in another clinical trial within 2 months prior to the start of the trial medication or during the trial period.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2006-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

REFERENCES:
- [Result] Sordal T, Grob P, Verhoeven C. Effects on bone mineral density of a monophasic combined oral contraceptive containing nomegestrol acetate/17beta-estradiol in comparison to levonorgestrel/ethinylestradiol. Acta Obstet Gynecol Scand. 2012 Nov;91(11):1279-85. doi: 10.1111/j.1600-0412.2012.01498.x. Epub 2012 Aug 21. PMID 22762147

RESULTS

PARTICIPANT FLOW:
Groups:
- NOMAC-E2: Monophasic combined oral contraceptive (COC) tablets containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-24, active tablets; Days 25-28, placebo tablets) for 26 consecutive 28-day cycles (2 years).
- LNG-EE: Monophasic combined oral contraceptive (COC) tablets containing 0.150 mg levonorgestrel (LNG) and 0.030 mg ethinylestradiol (EE) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-21, active tablets; Days 22-28, placebo tablets) for 26 consecutive 28-day cycles (2 years).
Period: Overall Study
Arm/Group | NOMAC-E2 | LNG-EE
Started | 56 | 54
Completed | 43 | 32
Not Completed | 13 | 22
Not completed — Unacceptable vaginal bleeding | 2 | 1
Not completed — Other Adverse Event (AE)/ Serious AE | 8 | 12
Not completed — Pregnancy | 0 | 1
Not completed — Pregnancy wish | 0 | 1
Not completed — Lost to Follow-up | 1 | 5
Not completed — Other Reason | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NOMAC-E2 | LNG-EE | Total
Number analyzed (Participants) | 56 | 54 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.0 (3.2) | 22.1 (2.0) | 22.6 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 54 | 110
  Male | 0 | 0 | 0
Baseline Z-scores of the Lumbar Spine (L2-L4) and Femoral Neck [Mean (Full Range); unit: score on a scale] — The Z-score measures the distance of the measured Bone Mineral Density (BMD) value from the appropriate normal age matched population mean value in units of standard deviation of this population. The following formula was used:
  Z-score= BMD value minus mean (age-matched reference population)/ SD (age-matched reference population).
  More negative scores indicate less BMD compared to age matched population, and more positive scores indicate higher BMD compared to age matched population.
  score on a scale
    Lumbar Spine | 0.351 [-2.30 to 2.70] | -0.106 [-2.19 to 2.88] | 0.127 [-2.30 to 2.88]
    Femoral Neck | 0.321 [-1.80 to 2.54] | 0.035 [-2.44 to 2.20] | 0.181 [-2.44 to 2.54]

OUTCOME MEASURES:

1. Secondary Outcome: Number of In-treatment Pregnancies (With +2 Day Window) Per 100 Woman Years of Exposure (Pearl Index)
Description: Contraceptive efficacy parameter of this trial was the Pearl Index. In-treatment pregnancies were pregnancies with an estimated date of conception from
  the day of first intake of trial medication up to and including the day of last(active or placebo) intake of trial medication extended with a maximum of two days. Each 13 cycles (28 days per cycle) of exposure constitutes a woman year. The Pearl Index was obtained by dividing the number of in-treatment pregnancies that occurred by the time (in 100 women years) that the women were under risk of becoming pregnant.
Time Frame: 2 years (26 cycles)
Population: Restricted Intent-To-Treat (ITT) analysis set included all participants treated, and further excluded non-pregnant participants without at least one cycle expected to be at risk for pregnancy(with recorded use of condoms or without confirmed sexual intercourse, as determined from the electronic diary data).
Measure: Number (95% Confidence Interval); unit: Pregnancies per 100 woman years
Units Other Than Participants: Woman years (rounded to nearest integer)
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 54 | 48
Number analyzed (Woman years (rounded to nearest integer)) | 72 | 58
Pregnancies per 100 woman years | 0.000 [0 to 5.1276] | 1.734 [0.0439 to 9.6621]

2. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Bleeding/ Spotting
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary cards. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough bleeding/spotting was defined as any episode that occurred during the "expected non-bleeding period" that was neither an early nor a continued withdrawal bleeding. Expected non-bleeding period: LNG-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 26 cycles (2 years total)
Population: The ITT group consisted of all participants who were treated; ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n= Number of participants with evaluable cycles.
Measure: Number; unit: participants
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 52
participants
  Cycle 1 (n=53 Nomac-E2/ n=52 LNG-EE) | 22 | 14
  Cycle 2 (n=53 Nomac-E2/ n=49 LNG-EE) | 12 | 6
  Cycle 3 (n=55 Nomac-E2/ n=48 LNG-EE) | 15 | 3
  Cycle 4 (n=53 Nomac-E2/ n=44 LNG-EE) | 12 | 2
  Cycle 5 (n=50 Nomac-E2/ n=44 LNG-EE) | 11 | 2
  Cycle 6 (n=51 Nomac-E2/ n=44 LNG-EE) | 10 | 5
  Cycle 7 (n=48 Nomac-E2/ n=42 LNG-EE) | 6 | 5
  Cycle 8 (n=47 Nomac-E2/ n=41 LNG-EE) | 4 | 3
  Cycle 9 (n=47 Nomac-E2/ n=40 LNG-EE) | 9 | 8
  Cycle 10 (n=45 Nomac-E2/ n=40 LNG-EE) | 7 | 1
  Cycle 11 (n=44 Nomac-E2/ n=40 LNG-EE) | 6 | 3
  Cycle 12 (n=42 Nomac-E2/ n=40 LNG-EE) | 5 | 4
  Cycle 13 (n=41 Nomac-E2/ n=39 LNG-EE) | 6 | 4
  Cycle 14 (n=42 Nomac-E2/ n=39 LNG-EE) | 3 | 3
  Cycle 15 (n=43 Nomac-E2/ n=38 LNG-EE) | 2 | 2
  Cycle 16 (n=43 Nomac-E2/ n=38 LNG-EE) | 6 | 2
  Cycle 17 (n=43 Nomac-E2/ n=37 LNG-EE) | 4 | 2
  Cycle 18 (n=43 Nomac-E2/ n=37 LNG-EE) | 1 | 3
  Cycle 19 (n=43 Nomac-E2/ n=37 LNG-EE) | 2 | 2
  Cycle 20 (n=42 Nomac-E2/ n=36 LNG-EE) | 4 | 2
  Cycle 21 (n=41 Nomac-E2/ n=35 LNG-EE) | 4 | 1
  Cycle 22 (n=42 Nomac-E2/ n=34 LNG-EE) | 2 | 1
  Cycle 23 (n=43 Nomac-E2/ n=35 LNG-EE) | 4 | 5
  Cycle 24 (n=43 Nomac-E2/ n=35 LNG-EE) | 2 | 3
  Cycle 25 (n=42 Nomac-E2/ n=33 LNG-EE) | 6 | 2
  Cycle 26 (n=32 Nomac-E2/ n=21 LNG-EE) | 3 | 0

3. Primary Outcome: Mean Change From Baseline in Z-scores of the Lumbar Spine (L2-L4) and Femoral Neck
Description: BMD was measured by a Dual Energy X-ray Absorptiometry (DEXA) machine. The Z-score measures the distance of the measured BMD value from the appropriate normal age matched population mean value in units of standard deviation of this population. More negative scores indicate less BMD compared to age matched population, & more positive scores indicate higher BMD compared to age matched population. The adjusted mean change from baseline to the after Cycle 26 visit of the Z-scores is estimated using a baseline-adjusted analysis of covariance (ANCOVA).
Time Frame: Baseline and after cycle 26 (2 years)
Population: All-Subjects-Treated (AST) group consisted of all randomized participants who took at least one dose of trial medication. The number of participants in the AST group with a baseline value and a Week 26 value is presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 54
score on a scale
  Lumbar Spine (n=42/ n=34) | 0.019 (0.242) [-0.049 to 0.108] | 0.121 (0.269) [0.020 to 0.195]
  Femoral Neck (n=42/ n=34 ) | -0.007 (0.228) [-0.068 to 0.073] | 0.044 (0.253) [-0.045 to 0.111]
Statistical Analysis 1: Comparison: NOMAC-E2 vs LNG-EE; Test type: Superiority or Other; p = 0.19, ANCOVA — No corrections for multiple comparisons were made for these safety parameters. The a-priori threshold for statistical significance was 0.05; The ANCOVA included the Z-score values at baseline as adjusted factor; Difference of adjusted means = -0.078, 95% CI 2-sided [-0.198 to 0.041] — NOMAC-E2 minus LNG-EE for lumbar spine (L2-L4)
Statistical Analysis 2: Comparison: NOMAC-E2 vs LNG-EE; Test type: Superiority or Other; p = 0.57, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The ANCOVA included the Z-score values at baseline as adjusted factor; Difference of adjusted means = -0.030, 95% CI 2-sided [-0.136 to 0.075] — NOMAC-E2 minus LNG-EE for femoral neck

4. Secondary Outcome: Number of Participants With an Occurrence of Absence of Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary cards. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Absence of withdrawal bleeding was defined as no bleeding/spotting episode that began during or continued into the "expected bleeding period". Expected bleeding period: LNG-EE group: 7-day period starting on Day 22 of the cycle; NOMAC-E2 group: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle.
Time Frame: Every 28-day cycle for 26 cycles (2 years total)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 52
participants
  Cycle 1 (n=53 Nomac-E2/ n=52 LNG-EE) | 4 | 2
  Cycle 2 (n=53 Nomac-E2/ n=49 LNG-EE) | 9 | 2
  Cycle 3 (n=55 Nomac-E2/ n=48 LNG-EE) | 9 | 1
  Cycle 4 (n=53 Nomac-E2/ n=44 LNG-EE) | 16 | 0
  Cycle 5 (n=50 Nomac-E2/ n=44 LNG-EE) | 10 | 0
  Cycle 6 (n=51 Nomac-E2/ n=44 LNG-EE) | 14 | 0
  Cycle 7 (n=48 Nomac-E2/ n=42 LNG-EE) | 15 | 1
  Cycle 8 (n=47 Nomac-E2/ n=41 LNG-EE) | 12 | 0
  Cycle 9 (n=47 Nomac-E2/ n=40 LNG-EE) | 13 | 3
  Cycle 10 (n=45 Nomac-E2/ n=40 LNG-EE) | 14 | 1
  Cycle 11 (n=44 Nomac-E2/ n=40 LNG-EE) | 16 | 0
  Cycle 12 (n=42 Nomac-E2/ n=40 LNG-EE) | 12 | 0
  Cycle 13 (n=41 Nomac-E2/ n=39 LNG-EE) | 11 | 0
  Cycle 14 (n=42 Nomac-E2/ n=39 LNG-EE) | 12 | 2
  Cycle 15 (n=43 Nomac-E2/ n=38 LNG-EE) | 21 | 2
  Cycle 16 (n=43 Nomac-E2/ n=38 LNG-EE) | 17 | 1
  Cycle 17 (n=43 Nomac-E2/ n=37 LNG-EE) | 18 | 1
  Cycle 18 (n=43 Nomac-E2/ n=37 LNG-EE) | 13 | 3
  Cycle 19 (n=43 Nomac-E2/ n=37 LNG-EE) | 18 | 2
  Cycle 20 (n=42 Nomac-E2/ n=36 LNG-EE) | 20 | 2
  Cycle 21 (n=41 Nomac-E2/ n=35 LNG-EE) | 17 | 2
  Cycle 22 (n=42 Nomac-E2/ n=34 LNG-EE) | 16 | 2
  Cycle 23 (n=43 Nomac-E2/ n=35 LNG-EE) | 17 | 4
  Cycle 24 (n=43 Nomac-E2/ n=35 LNG-EE) | 19 | 3
  Cycle 25 (n=42 Nomac-E2/ n=33 LNG-EE) | 15 | 2
  Cycle 26 (n=32 Nomac-E2/ n=21 LNG-EE) | 24 | 11

5. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary cards. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough bleeding was defined as any bleeding episode that occurred during the "expected non-bleeding period" that was neither part of an early nor continued withdrawal bleeding. Expected non-bleeding period: LNG-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 26 cycles (2 years total)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 52
participants
  Cycle 1 (n=53 Nomac-E2/ n=52 LNG-EE) | 6 | 1
  Cycle 2 (n=53 Nomac-E2/ n=49 LNG-EE) | 2 | 1
  Cycle 3 (n=55 Nomac-E2/ n=48 LNG-EE) | 2 | 1
  Cycle 4 (n=53 Nomac-E2/ n=44 LNG-EE) | 3 | 0
  Cycle 5 (n=50 Nomac-E2/ n=44 LNG-EE) | 2 | 1
  Cycle 6 (n=51 Nomac-E2/ n=44 LNG-EE) | 1 | 1
  Cycle 7 (n=48 Nomac-E2/ n=42 LNG-EE) | 0 | 1
  Cycle 8 (n=47 Nomac-E2/ n=41 LNG-EE) | 1 | 1
  Cycle 9 (n=47 Nomac-E2/ n=40 LNG-EE) | 2 | 0
  Cycle 10 (n=45 Nomac-E2/ n=40 LNG-EE) | 1 | 0
  Cycle 11 (n=44 Nomac-E2/ n=40 LNG-EE) | 1 | 1
  Cycle 12 (n=42 Nomac-E2/ n=40 LNG-EE) | 1 | 1
  Cycle 13 (n=41 Nomac-E2/ n=39 LNG-EE) | 2 | 1
  Cycle 14 (n=42 Nomac-E2/ n=39 LNG-EE) | 1 | 1
  Cycle 15 (n=43 Nomac-E2/ n=38 LNG-EE) | 1 | 1
  Cycle 16 (n=43 Nomac-E2/ n=38 LNG-EE) | 1 | 0
  Cycle 17 (n=43 Nomac-E2/ n=37 LNG-EE) | 2 | 0
  Cycle 18 (n=43 Nomac-E2/ n=37 LNG-EE) | 0 | 0
  Cycle 19 (n=43 Nomac-E2/ n=37 LNG-EE) | 1 | 0
  Cycle 20 (n=42 Nomac-E2/ n=36 LNG-EE) | 2 | 0
  Cycle 21 (n=41 Nomac-E2/ n=35 LNG-EE) | 1 | 0
  Cycle 22 (n=42 Nomac-E2/ n=34 LNG-EE) | 0 | 0
  Cycle 23 (n=43 Nomac-E2/ n=35 LNG-EE) | 1 | 1
  Cycle 24 (n=43 Nomac-E2/ n=35 LNG-EE) | 0 | 1
  Cycle 25 (n=42 Nomac-E2/ n=33 LNG-EE) | 0 | 0
  Cycle 26 (n=32 Nomac-E2/ n=21 LNG-EE) | 0 | 0

6. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Spotting (Spotting Only)
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary cards. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough spotting was defined as any spotting episode that occurred during the "expected non-bleeding period" that was neither part of an early nor continued withdrawal bleeding. Expected non-bleeding period: LNG-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 26 cycles (2 years total)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 52
participants
  Cycle 1 (n=53 Nomac-E2/ n=52 LNG-EE) | 17 | 13
  Cycle 2 (n=53 Nomac-E2/ n=49 LNG-EE) | 10 | 5
  Cycle 3 (n=55 Nomac-E2/ n=48 LNG-EE) | 14 | 2
  Cycle 4 (n=53 Nomac-E2/ n=44 LNG-EE) | 9 | 2
  Cycle 5 (n=50 Nomac-E2/ n=44 LNG-EE) | 11 | 1
  Cycle 6 (n=51 Nomac-E2/ n=44 LNG-EE) | 9 | 4
  Cycle 7 (n=48 Nomac-E2/ n=42 LNG-EE) | 6 | 4
  Cycle 8 (n=47 Nomac-E2/ n=41 LNG-EE) | 3 | 2
  Cycle 9 (n=47 Nomac-E2/ n=40 LNG-EE) | 8 | 8
  Cycle 10 (n=45 Nomac-E2/ n=40 LNG-EE) | 6 | 1
  Cycle 11 (n=44 Nomac-E2/ n=40 LNG-EE) | 6 | 3
  Cycle 12 (n=42 Nomac-E2/ n=40 LNG-EE) | 4 | 3
  Cycle 13 (n=41 Nomac-E2/ n=39 LNG-EE) | 5 | 3
  Cycle 14 (n=42 Nomac-E2/ n=39 LNG-EE) | 2 | 2
  Cycle 15 (n=43 Nomac-E2/ n=38 LNG-EE) | 1 | 2
  Cycle 16 (n=43 Nomac-E2/ n=38 LNG-EE) | 5 | 2
  Cycle 17 (n=43 Nomac-E2/ n=37 LNG-EE) | 2 | 2
  Cycle 18 (n=43 Nomac-E2/ n=37 LNG-EE) | 1 | 3
  Cycle 19 (n=43 Nomac-E2/ n=37 LNG-EE) | 1 | 2
  Cycle 20 (n=42 Nomac-E2/ n=36 LNG-EE) | 2 | 2
  Cycle 21 (n=41 Nomac-E2/ n=35 LNG-EE) | 3 | 1
  Cycle 22 (n=42 Nomac-E2/ n=34 LNG-EE) | 2 | 1
  Cycle 23 (n=43 Nomac-E2/ n=35 LNG-EE) | 4 | 4
  Cycle 24 (n=43 Nomac-E2/ n=35 LNG-EE) | 2 | 2
  Cycle 25 (n=42 Nomac-E2/ n=33 LNG-EE) | 6 | 2
  Cycle 26 (n=32 Nomac-E2/ n=21 LNG-EE) | 3 | 0

7. Secondary Outcome: Number of Participants With an Occurrence of Early Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary cards. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Early withdrawal bleeding was defined as any withdrawal bleeding that started before the current "expected bleeding period". Expected bleeding period: LNG-EE group: 7-day period starting on Day 22 of the cycle; NOMAC-E2 group: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle.
Time Frame: Every 28-day cycle for 26 cycles (2 years total)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 52
participants
  Cycle 1 (n=53 Nomac-E2/ n=52 LNG-EE) | 5 | 7
  Cycle 2 (n=53 Nomac-E2/ n=49 LNG-EE) | 3 | 4
  Cycle 3 (n=55 Nomac-E2/ n=48 LNG-EE) | 3 | 3
  Cycle 4 (n=53 Nomac-E2/ n=44 LNG-EE) | 1 | 4
  Cycle 5 (n=50 Nomac-E2/ n=44 LNG-EE) | 3 | 3
  Cycle 6 (n=51 Nomac-E2/ n=44 LNG-EE) | 1 | 3
  Cycle 7 (n=48 Nomac-E2/ n=42 LNG-EE) | 4 | 4
  Cycle 8 (n=47 Nomac-E2/ n=41 LNG-EE) | 1 | 3
  Cycle 9 (n=47 Nomac-E2/ n=40 LNG-EE) | 0 | 3
  Cycle 10 (n=45 Nomac-E2/ n=40 LNG-EE) | 1 | 4
  Cycle 11 (n=44 Nomac-E2/ n=40 LNG-EE) | 1 | 3
  Cycle 12 (n=42 Nomac-E2/ n=40 LNG-EE) | 2 | 3
  Cycle 13 (n=41 Nomac-E2/ n=39 LNG-EE) | 1 | 2
  Cycle 14 (n=42 Nomac-E2/ n=39 LNG-EE) | 0 | 0
  Cycle 15 (n=43 Nomac-E2/ n=38 LNG-EE) | 0 | 1
  Cycle 16 (n=43 Nomac-E2/ n=38 LNG-EE) | 0 | 2
  Cycle 17 (n=43 Nomac-E2/ n=37 LNG-EE) | 0 | 0
  Cycle 18 (n=43 Nomac-E2/ n=37 LNG-EE) | 0 | 0
  Cycle 19 (n=43 Nomac-E2/ n=37 LNG-EE) | 0 | 1
  Cycle 20 (n=42 Nomac-E2/ n=36 LNG-EE) | 0 | 1
  Cycle 21 (n=41 Nomac-E2/ n=35 LNG-EE) | 0 | 2
  Cycle 22 (n=42 Nomac-E2/ n=34 LNG-EE) | 1 | 2
  Cycle 23 (n=43 Nomac-E2/ n=35 LNG-EE) | 0 | 1
  Cycle 24 (n=43 Nomac-E2/ n=35 LNG-EE) | 0 | 1
  Cycle 25 (n=42 Nomac-E2/ n=33 LNG-EE) | 1 | 2
  Cycle 26 (n=32 Nomac-E2/ n=21 LNG-EE) | 1 | 0

8. Secondary Outcome: Number of Participants With an Occurrence of Continued Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary cards. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Continued withdrawal bleeding was defined as any withdrawal bleeding that continued into the "expected non-bleeding period" of the next cycle. Expected non-bleeding period: LNG-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 26 cycles (2 years total) including one week after stopping treatment
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 52
participants
  Cycle 1 (n=53 Nomac-E2/ n=52 LNG-EE) | 10 | 24
  Cycle 2 (n=53 Nomac-E2/ n=49 LNG-EE) | 14 | 19
  Cycle 3 (n=53 Nomac-E2/ n=45 LNG-EE) | 14 | 17
  Cycle 4 (n=51 Nomac-E2/ n=43 LNG-EE) | 9 | 19
  Cycle 5 (n=50 Nomac-E2/ n=44 LNG-EE) | 9 | 18
  Cycle 6 (n=50 Nomac-E2/ n=43 LNG-EE) | 11 | 14
  Cycle 7 (n=48 Nomac-E2/ n=41 LNG-EE) | 7 | 15
  Cycle 8 (n=47 Nomac-E2/ n=41 LNG-EE) | 10 | 16
  Cycle 9 (n=47 Nomac-E2/ n=40 LNG-EE) | 11 | 9
  Cycle 10 (n=44 Nomac-E2/ n=39 LNG-EE) | 5 | 13
  Cycle 11 (n=43 Nomac-E2/ n=40 LNG-EE) | 5 | 16
  Cycle 12 (n=42 Nomac-E2/ n=40 LNG-EE) | 6 | 18
  Cycle 13 (n=41 Nomac-E2/ n=38 LNG-EE) | 8 | 9
  Cycle 14 (n=42 Nomac-E2/ n=38 LNG-EE) | 10 | 12
  Cycle 15 (n=43 Nomac-E2/ n=38 LNG-EE) | 6 | 10
  Cycle 16 (n=43 Nomac-E2/ n=38 LNG-EE) | 4 | 11
  Cycle 17 (n=43 Nomac-E2/ n=37 LNG-EE) | 6 | 14
  Cycle 18 (n=43 Nomac-E2/ n=37 LNG-EE) | 4 | 14
  Cycle 19 (n=43 Nomac-E2/ n=36 LNG-EE) | 7 | 15
  Cycle 20 (n=42 Nomac-E2/ n=36 LNG-EE) | 3 | 13
  Cycle 21 (n=41 Nomac-E2/ n=34 LNG-EE) | 6 | 16
  Cycle 22 (n=42 Nomac-E2/ n=34 LNG-EE) | 7 | 13
  Cycle 23 (n=43 Nomac-E2/ n=35 LNG-EE) | 4 | 12
  Cycle 24 (n=43 Nomac-E2/ n=35 LNG-EE) | 3 | 10
  Cycle 25 (n=42 Nomac-E2/ n=33 LNG-EE) | 3 | 7
  Cycle 26 (n=4Nomac-E2/ n=1 LNG-EE) | 0 | 0

9. Secondary Outcome: Average Number of Breakthrough Bleeding-Spotting Days
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary cards. Participants documented whether vaginal bleeding was present, and if so, indicated whether it was considered to be spotting or bleeding. Breakthrough bleeding/spotting was defined as any bleeding/spotting episode that occurred during the "expected non-bleeding period" that was neither an early nor a continued withdrawal bleeding. Expected non-bleeding period: LNG-EE: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 26 cycles (2 years total)
Population: ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n= number of participants who had breakthrough bleeding/spotting for the respective cycle.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 52
days
  Cycle 1 (n=22 Nomac-E2/ n=14 LNG-EE) | 4.1 (3.1) | 2.2 (1.9)
  Cycle 2 (n=12 Nomac-E2/ n=6 LNG-EE) | 3.8 (3.1) | 4.8 (1.9)
  Cycle 3 (n=15 Nomac-E2/ n=3 LNG-EE) | 4.1 (3.8) | 4.0 (1.7)
  Cycle 4 (n=12 Nomac-E2/ n=2 LNG-EE) | 4.0 (2.8) | 1.5 (0.7)
  Cycle 5 (n=11 Nomac-E2/ n=2 LNG-EE) | 3.7 (2.3) | 6.5 (6.4)
  Cycle 6 (n=10 Nomac-E2/ n=5 LNG-EE) | 2.0 (1.2) | 2.6 (1.8)
  Cycle 7 (n=6 Nomac-E2/ n=5 LNG-EE) | 3.0 (1.9) | 2.6 (0.9)
  Cycle 8 (n=4 Nomac-E2/ n=3 LNG-EE) | 2.3 (1.5) | 2.0 (1.0)
  Cycle 9 (n=9 Nomac-E2/ n=8 LNG-EE) | 2.2 (1.4) | 2.1 (1.0)
  Cycle 10 (n=7 Nomac-E2/ n=1 LNG-EE) | 2.0 (0.8) | 2.0 (NA) — Value for one participant, therefore, standard deviation does not apply.
  Cycle 11 (n=6 Nomac-E2/ n=3 LNG-EE) | 2.0 (1.1) | 2.3 (1.2)
  Cycle 12 (n=5 Nomac-E2/ n=4 LNG-EE) | 3.2 (0.8) | 4.0 (2.4)
  Cycle 13 (n=6 Nomac-E2/ n=4 LNG-EE) | 3.0 (2.1) | 3.0 (2.2)
  Cycle 14 (n=3 Nomac-E2/ n=3 LNG-EE) | 1.3 (0.6) | 2.7 (1.5)
  Cycle 15 (n=2 Nomac-E2/ n=2 LNG-EE) | 2.0 (1.4) | 7.5 (2.1)
  Cycle 16 (n=6 Nomac-E2/ n=2 LNG-EE) | 1.5 (0.5) | 1.5 (0.7)
  Cycle 17 (n=4 Nomac-E2/ n=2 LNG-EE) | 1.8 (1.0) | 2.0 (1.4)
  Cycle 18 (n=1 Nomac-E2/ n=3 LNG-EE) | 3.0 (NA) — Value for one participant, therefore, standard deviation does not apply. | 3.0 (2.0)
  Cycle 19 (n=2 Nomac-E2/ n=2 LNG-EE) | 2.0 (1.4) | 6.0 (1.4)
  Cycle 20 (n=4 Nomac-E2/ n=2 LNG-EE) | 3.5 (2.1) | 4.0 (4.2)
  Cycle 21 (n=4 Nomac-E2/ n=1 LNG-EE) | 2.3 (1.3) | 5.0 (NA) — Value for one participant, therefore, standard deviation does not apply.
  Cycle 22 (n=2 Nomac-E2/ n=1 LNG-EE) | 3.0 (1.4) | 6.0 (NA) — Value for one participant, therefore, standard deviation does not apply.
  Cycle 23 (n=4 Nomac-E2/ n=5 LNG-EE) | 3.8 (2.9) | 3.4 (1.8)
  Cycle 24 (n=2 Nomac-E2/ n=3 LNG-EE) | 2.0 (1.4) | 4.7 (3.2)
  Cycle 25 (n=6 Nomac-E2/ n=2 LNG-EE) | 2.2 (1.3) | 3.5 (3.5)
  Cycle 26 (n=3 Nomac-E2/ n=0 LNG-EE) | 2.3 (2.3) | NA (NA) — Mean and Standard Deviation does not apply for 0 participants.

10. Secondary Outcome: Average Number of Withdrawal Bleeding-spotting Days
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary cards. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Withdrawal bleeding was defined as bleeding/spotting episode that started during or continued into the "expected bleeding period". Expected bleeding period: LNG-EE group: 7-day period starting on Day 22 of the cycle; NOMAC-E2 group: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle.
Time Frame: Every 28-day cycle for 26 cycles (2 years total)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NOMAC-E2 | LNG-EE
Number analyzed (Participants) | 56 | 52
days
  Cycle 1 (n=49 Nomac-E2/ n=50 LNG-EE) | 4.7 (2.7) | 6.7 (4.0)
  Cycle 2 (n=44 Nomac-E2/ n=47 LNG-EE) | 4.7 (2.1) | 5.3 (1.8)
  Cycle 3 (n=46 Nomac-E2/ n=47 LNG-EE) | 4.4 (2.0) | 5.2 (1.6)
  Cycle 4 (n=37 Nomac-E2/ n=44 LNG-EE) | 4.3 (2.0) | 5.5 (2.1)
  Cycle 5 (n=40 Nomac-E2/ n=44 LNG-EE) | 4.1 (2.7) | 5.6 (2.9)
  Cycle 6 (n=37 Nomac-E2/ n=44 LNG-EE) | 4.0 (1.7) | 5.0 (1.5)
  Cycle 7 (n=33 Nomac-E2/ n=41 LNG-EE) | 4.0 (1.8) | 5.1 (1.6)
  Cycle 8 (n=35 Nomac-E2/ n=41 LNG-EE) | 3.5 (1.5) | 5.1 (1.5)
  Cycle 9 (n=34 Nomac-E2/ n=37 LNG-EE) | 3.6 (1.3) | 5.4 (2.5)
  Cycle 10 (n=31 Nomac-E2/ n=39 LNG-EE) | 3.5 (1.2) | 5.4 (2.4)
  Cycle 11 (n=28 Nomac-E2/ n=40 LNG-EE) | 3.9 (1.5) | 5.1 (1.5)
  Cycle 12 (n=30 Nomac-E2/ n=40 LNG-EE) | 3.8 (1.9) | 5.1 (1.5)
  Cycle 13 (n=30 Nomac-E2/ n=39 LNG-EE) | 3.4 (1.5) | 4.8 (1.8)
  Cycle 14 (n=30 Nomac-E2/ n=37 LNG-EE) | 3.8 (1.6) | 4.9 (1.2)
  Cycle 15 (n=22 Nomac-E2/ n=36 LNG-EE) | 3.6 (1.6) | 4.8 (1.2)
  Cycle 16 (n=26 Nomac-E2/ n=37 LNG-EE) | 3.2 (1.1) | 4.9 (2.1)
  Cycle 17 (n=25 Nomac-E2/ n=36 LNG-EE) | 4.0 (1.9) | 4.6 (1.3)
  Cycle 18 (n=30 Nomac-E2/ n=34 LNG-EE) | 3.2 (1.3) | 4.8 (1.3)
  Cycle 19 (n=25 Nomac-E2/ n=35 LNG-EE) | 3.7 (1.5) | 4.9 (1.6)
  Cycle 20 (n=22 Nomac-E2/ n=34 LNG-EE) | 3.4 (1.2) | 5.0 (1.4)
  Cycle 21 (n=24 Nomac-E2/ n=33 LNG-EE) | 3.4 (1.8) | 4.8 (1.6)
  Cycle 22 (n=26 Nomac-E2/ n=32 LNG-EE) | 3.7 (1.5) | 5.1 (1.9)
  Cycle 23 (n=26 Nomac-E2/ n=31 LNG-EE) | 3.5 (1.6) | 5.0 (1.4)
  Cycle 24 (n=24 Nomac-E2/ n=32 LNG-EE) | 3.7 (2.2) | 4.9 (1.5)
  Cycle 25 (n=27 Nomac-E2/ n=31 LNG-EE) | 3.4 (2.0) | 5.2 (3.2)
  Cycle 26 (n=8 Nomac-E2/ n=10 LNG-EE) | 3.1 (1.4) | 4.2 (0.6)

ADVERSE EVENTS:
Arm/Group | NOMAC-E2 | LNG-EE
Serious Adverse Events (participants affected / at risk) | 1/56 | 1/54
Other Adverse Events (participants affected / at risk) | 42/56 | 43/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOMAC-E2 (N=56) | LNG-EE (N=54)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOMAC-E2 (N=56) | LNG-EE (N=54)
Palpitations (Cardiac disorders) | 3 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Chlamydial cervicitis (Infections and infestations) | 0 (0) | 3 (4)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (4)
Influenza (Infections and infestations) | 10 (13) | 9 (11)
Nasopharyngitis (Infections and infestations) | 17 (26) | 18 (28)
Sinusitis (Infections and infestations) | 2 (2) | 3 (4)
Vaginitis bacterial (Infections and infestations) | 0 (0) | 3 (3)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (3) | 4 (4)
Weight increased (Investigations) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 7 (15)
Libido decreased (Psychiatric disorders) | 3 (3) | 0 (0)
Mood altered (Psychiatric disorders) | 6 (6) | 6 (6)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Dyspareunia (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hot flush (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR recognizes the right of the investigator(s) to publish, but all publications must be based on data validated and released by the SPONSOR. Any such scientific paper, presentation, or other communication concerning the clinical trial will first be submitted to the SPONSOR, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.